CLINICAL TRIAL: NCT02036671
Title: Novel Endovascular Access Trial (NEAT): A Study of the FLEX System for Percutaneous AV Fistula Creation in Hemodialysis Patients
Brief Title: Novel Endovascular Access Trial (NEAT)
Acronym: NEAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VAP-0001
Record Dates: First submitted 2014-01-10; First posted 2014-01-15 (Estimated); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Chronic Kidney Disease
Keywords: Arteriovenous fistula; Fistula; Chronic kidney disease; Percutaneous; Kidney Disease; Kidney Failure, Chronic; Urologic Diseases; Renal Insufficiency, Chronic; Renal Insufficiency; CKD; hemodialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Arteriovenous Fistula; Fistula; Kidney Diseases; Kidney Failure, Chronic; Urologic Diseases; Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EndoAVF (Experimental): The FLEX System will be used to percutaneously create a fistula in CKD patients who require hemodialysis vascular access
  Interventions: Device: The FLEX System will be used to percutaneously create a fistula in CKD patients who require hemodialysis vascular access

INTERVENTIONS:
Device: The FLEX System will be used to percutaneously create a fistula in CKD patients who require hemodialysis vascular access

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of the FLEX System when used to create an arteriovenous fistula (AVF or AV fistula) percutaneously in patients with Chronic Kidney Disease (CKD) who require hemodialysis vascular access.

DETAILED DESCRIPTION:
This is a 12 month multi-center non-randomized investigational study to evaluate the safety and efficacy of the FLEX system to create an endovascular AVF in patients with CKD who require hemodialysis vascular access.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for a native surgical arteriovenous fistula, as determined by the treating physician.
* Adult (age >18 years old).
* Established, non-reversible kidney failure requiring hemodialysis.
* Written informed consent obtained.

Exclusion Criteria:

* Functioning surgical access in the planned treatment arm.
* Pregnant women.
* New York Heart Association (NYHA) class III or IV heart failure.
* Allergy to contrast dye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint: | within 3 months
  The percentage of patients with fistula maturation/usability defined as endoAVF that is free of stenosis or thrombosis, with brachial artery flow of at least 500 ml/min and at least 4 mm vein diameter (as measured by duplex ultrasound) OR patient was dialyzed using 2 needles.

SECONDARY OUTCOMES:
Safety Endpoint | within 3 months
  The percentage of patients who experience one or more serious study device related adverse events during the first 3 months following AVF creation
EndoAVF-related Re-intervention Rate | 3, 6 and 12 months
  The re-intervention rate for endoAVF (defined as any intervention required to maintain or re-establish patency) will be calculated at 3, 6 and 12 months post index procedure.
Primary Patency | 3, 6 and 12 months
  Time from successful endoAVF creation to the first intervention designed to address thrombosis or stenosis, assist in maturation or cannulation of endoAVF, or endoAVF abandonment.
Cumulative Patency | 3, 6 and 12 months
  Time from creation to the abandonment of endoAVF (censor patients with renal transplant)
Functional Usability | 4 weeks post procedure, up to 12 months
  2-needle cannulation of the endoAVF for prescribed dialysis in ≥ 2/3 of dialysis sessions over a 4 consecutive week period within 12 months of endoAVF creation.

CONTACTS AND LOCATIONS:
Overall Officials: Charmaine Lok, MD, MSC, FRCPC, Principal Investigator — The Toronto General Hospital; Dheeraj Rajan, MD, BSc, FRCPC, FSIR, Principal Investigator — The Toronto General Hospital
Locations (9):
- Australia (2):
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Alfred Hospital, Melbourne, Victoria
- Canada (6):
  - St. Paul's Hospital, Vancouver, British Columbia
  - QE II Health Sciences Center, Halifax, Nova Scotia
  - London Health Sciences Centre, London, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - The Toronto General Hospital, Toronto, Ontario
  - CHUM, Notre-Dame Hospital, Montreal, Quebec
- Auckland City Hospital, Grafton, New Zealand